CLINICAL TRIAL: NCT02612324
Title: An Evaluation of Pono Choices: A Culturally Responsive Teen Pregnancy and STI Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: IMPAQ International, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TP2AH000017
Record Dates: First submitted 2015-11-12; First posted 2015-11-23 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Teen Pregnancy; Sexually Transmitted Infections
Keywords: adolescents; teen pregnancy prevention; sexually transmitted infections prevention; place-based programs; health education
MeSH Terms: conditions — Sexually Transmitted Diseases; Health Education | interventions — Commerce

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pono Choices (Experimental): Pono Choices: A Culturally Responsive Teen Pregnancy and STI Prevention Program for Middle School Youth in Hawaii. The program includes 9.5 hours of scripted lessons or modules.
  Interventions: Behavioral: Pono Choices
- Business as Usual (Active Comparator): Middle school sexual health content or programs chosen by control group schools.
  Interventions: Behavioral: Business as Usual

INTERVENTIONS:
Behavioral: Pono Choices — Medically accurate teen pregnancy and STI prevention education delivered through a place-based framework integrating Hawaiian cultural activities that draw upon both historical and local references.
  Arms: Pono Choices
Behavioral: Business as Usual — Teen pregnancy and STI prevention education left to the discretion of the school.
  Arms: Business as Usual

SUMMARY:
The purpose of this study is to determine the impact Pono Choices has among youth for teen pregnancy and STI prevention measures such as: initiation of sexual activity; engagement in high risk sexual behaviors; knowledge of pregnancy and STI prevention; attitudes toward healthy sexual behaviors; skills in managing relationships and choices; and intentions about future sexual activity.

DETAILED DESCRIPTION:
The study used a cluster randomized controlled design to evaluate the impact of Pono Choices. Thirty-six middle schools in Hawaii were randomly assigned to participate as either a treatment or control school. Treatment school teachers were trained to deliver Pono Choices. Control school teachers did not receive training and chose their own middle school sexual health education curricula.

Over 1,700 7th and 8th grade students in 34 Hawaii schools enrolled into the study. As part of the study, students were invited to participate in baseline and follow-up surveys. The student survey responses were used to determine the impact Pono Choices has on teen pregnancy and STI prevention measures.

ELIGIBILITY:
Inclusion Criteria:

* Cluster level: Schools with grades 7 and 8 in Hawaii
* Person level: Students with parent consent and who read and understand English

Exclusion Criteria:

* Cluster level: Public middle schools which included grade 6
* Person level: Students who did not provide written assent

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1783 (Actual)
Dates: Start 2012-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Initiation of sexual activity assessed by the percent reporting on the questionnaire that they have had sexual intercourse. | 1 year

SECONDARY OUTCOMES:
Engagement in high risk sexual behaviors assessed by the percent reporting on the questionnaire that they have engaged in sexual intercourse without a condom or other effective method of birth control in the past 3 months. | 1 year

OTHER OUTCOMES:
Knowledge related to pregnancy & STI prevention assessed by the percent of pregnancy and STI prevention knowledge items on the questionnaire answered correctly. | 1 year
Attitudes related to teen pregnancy & STI prevention behaviors assessed by the average rating of scale items on the questionnaire on the importance of healthy sexual behaviors. | 1 year
Skills related to teen pregnancy & STI prevention assessed by the average rating of scale items on the questionnaire on difficulty of skills related to managing relationship and choices. | 1 year
Intentions to have sex assessed by the scale response on the questionnaire on intention to have sex in the next 12 months. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kelly D Roberts, PhD, Principal Investigator — University of Hawaii at Manoa

REFERENCES:
- [Background] Manaseri H, Uehara D, Roberts K. Making Pono Choices: a collaborative approach to developing a culturally responsive teen pregnancy and sexually transmitted infections prevention curriculum in Hawai'i. Matern Child Health J. 2014 Dec;18(10):2332-40. doi: 10.1007/s10995-013-1395-6. PMID 24293268
- [Background] Manaseri, H, Roberts, K, Stofocik, K, Manuel, N, Uehara, D (2014). Culture as a Protective Factor: The Use of Storytelling in a Teen Pregnancy and STI Prevention Curriculum. Health Care Current Reviews, 2(3). doi:dx.doi.org/10.4172/hccr.1000127
- [Result] Abe Y, Barker LT, Chan V, Eucogco J. Culturally Responsive Adolescent Pregnancy and Sexually Transmitted Infection Prevention Program for Middle School Students in Hawai'i. Am J Public Health. 2016 Sep;106(S1):S110-S116. doi: 10.2105/AJPH.2016.303395. PMID 27689477
- [Result] Manaseri H, Roberts KD, Barker LT, Tom T. Pono Choices: Lessons for School Leaders From the Evaluation of a Teen Pregnancy Prevention Program. J Sch Health. 2019 Apr;89(4):246-256. doi: 10.1111/josh.12733. Epub 2019 Feb 11. PMID 30740698
- See also: Pono Choices Project website (curriculum development page) — http://www.cds.hawaii.edu/ponochoices/facilitators/curriculum-development/
- See also: AMCHP Best Practice Award Implementation Guide for Pono Choices — http://www.amchp.org/programsandtopics/BestPractices/InnovationStation/ISDocs/Implementation%20Handout_Pono%20Choices%202019.pdf